CLINICAL TRIAL: NCT01271205
Title: Red Cell Distribution Width and Mortality in Adult Pneumonia Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Eyal Braun, MD, Rambam Health Care Campus
Other Study IDs: 580CTIL
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2010-12

CONDITIONS: Pneumonia
Keywords: pneumonia; RDW; mortality; prognostic factor
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Abstract Pneumonia is a leading cause of severe morbidity and mortality among adults. During the last two decades, several scores were developed to evaluate the probability of morbidity and mortality among patients with community acquired pneumonia (CAP), such as the PORT score and the CURB65. Recently, several studies showed that elevated Red Cell Distribution Width (RDW) could be used as a prognostic tool for predicting severe morbidity and mortality among patients with cardiac diseases.

RDW is a quantitative measure for red blood cell (RBC) size variability. Recent studies have suggested that high levels of RDW are in association with higher mortality among cardiovascular patients.

RDW has not yet been studied as a prognostic sign in CAP. The goal of this study is to examine the role of RDW as a prognostic factor for severe morbidity and mortality among patients who were hospitalized with CAP , independently to Hemoglobin levels, renal function and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

patients 18 years and older, hospitalized due to pneumonia between 2005-2010. All patients must have RDW values.

-

Exclusion Criteria:

* under 18 no RDW value The primary cause of hospitalization was not pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-01